CLINICAL TRIAL: NCT02280798
Title: Endometrial Gene Expression in Different Protocols of Endometrial Preparation
Brief Title: Endometrial Gene Expression in Different Protocols of Endometrial Preparation for Embryo Transfer'
Acronym: ERA
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Collaborators: Igenomix (Industry)
Responsible Party: Principal Investigator, mcerrillo, MD, IVI Madrid
Other Study IDs: 1407-MAD-056-MC
Record Dates: First submitted 2014-09-16; First posted 2014-11-03 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Endometrial
Keywords: ERA

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — endometrial biopsies for ADN analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pilot study: A total of 5 volunteers from our egg donation program were included in the study with 4 endometrial biopsies for each one after 4 diferente protocols
  * Endometrial biopsy after Stimulated cycle
  * Endometrial biopsy after Natural Cycle
  * Endometrial biopsy after Natural modified cycle: the biopsy is taken seven days after the hCG
  * Endometrial biopsy after Hormone Replacement Therapy Cycle
  Interventions: Procedure: Endometrial Biopsy

INTERVENTIONS:
Procedure: Endometrial Biopsy — 4 endometrial biopsy

SUMMARY:
Do differences in endometrial gene expression exist after different protocols of endometrial preparation for embryo transfer? The recent apparition of endometrial receptive arrays technology let us know if endometrial is receptive or not in patients with some problems of infertility as implantation failure, for that we want to know if this technology would tell us if the different kind of protocols for endometrial preparation origin differences that could explain some of the founded results.

DETAILED DESCRIPTION:
Do differences in endometrial gene expression exist after different protocols of endometrial preparation for embryo transfer? The clinical results in different publications showed different results, some of them described the natural cycle superior as the substituted cycles, and in contrast other large series showed superior results in substituted cycles than natural but with an increased of pregnancies losses. The recent apparition of endometrial receptive arrays technology let us know if endometrial is receptive or not in patients with some problems of infertility as implantation failure, for that we want to know if this technology would tell us if the different kind of protocols for endometrial preparation origin differences that could explain some of the founded results.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* regular menstrual cycles (between 25 and 35 days)
* normal basal hormones(follicle-stimulating hormone [FSH] and LH <10 IU/ mL and estradiol <60 pg/mL)
* normal karyotype
* body massindex between 18 and 25 kg/m2
* negative serology
* normal cervical cytology in the past year, and a vaginal ultrasound without evidence of any pathologic conditions

Exclusion Criteria:

* endometriosis
* polycystic ovariansyndrome
* use of an intrauterine device in the last 3 months.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 5 volunteers from our egg donation program were included in the study from Setember 2014 to jnuary 2015
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Endometrial receptivity | 4 months
  Total RNA was extracted using the TRIzol method according to the manufacturer's recommendations (Life Technologies). Approximately 1-2 mg of total RNA was obtained per milligram of endometrial tissue. The RNA quality was assessed by loading 300 ng of total RNA onto an RNA LabChip and was analyzed in an A2100 Bioanalyzer (Agilent Technologies). Only samples with a RNA integrity number >7 were selected for microarray analysis.
  Sample preparation and hybridization was adapted from the Agilent technical manual. Hybridized microarrays were scanned in an Axon 4100A scanner (Molecular Devices), and the data were extracted with the GenePix Pro 6.0 software (Molecular Devices). The ERA microarray validation has been previously published. Reverse transcriptase-polymerase chain reaction (PCR) was performed for four selected up-regulated genes: GPX3, FXYD2, SPP1, and MT1G.
  The ERA gene expression values were preprocessed, normalized, and statistically analyzed. Briefly, the half background

SECONDARY OUTCOMES:
Hormonal profile | LH,E2,P4
  Hormonal profile different dates of protocols

CONTACTS AND LOCATIONS:
Overall Officials: Cerrillo M Maria, doctor, Principal Investigator — IVI Madrid
Locations (1):
- Maria Cerrillo, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes